CLINICAL TRIAL: NCT05656742
Title: Effects of Vitamin D on Cardiovascular Health in Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Melissa Witman, Associate Professor, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1957713
Record Dates: First submitted 2022-11-10; First posted 2022-12-19 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Vitamin d Deficiency
Keywords: vitamin D; black women; blood pressure; sleep; vascular
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: All participants will receive the same intervention: 8 weeks of daily oral vitamin D3 supplements, each containing 5,000 IU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D (Experimental): 5,000 IU of oral vitamin D3 in white powder form, daily for 8 continuous weeks
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — oral vitamin D3

SUMMARY:
The goal of this clinical trial is to understand the effects of oral vitamin D3 supplementation on various cardiovascular risk factors in generally healthy, young adult black women who are vitamin D deficient or insufficient at baseline.

The main questions it aims to answer are:

* Does 8 weeks of oral vitamin D3 supplementation (5,000 IU per day) improve 24 hour blood pressure metrics in generally healthy, young adult black women who are vitamin D deficient or insufficient at baseline?
* Does 8 weeks of oral vitamin D3 supplementation (5,000 IU per day) improve subjective and objectively estimated sleep health metrics in generally healthy, young adult black women who are vitamin D deficient or insufficient at baseline?
* Does 8 weeks of oral vitamin D3 supplementation (5,000 IU per day) improve various measures of blood vessel structure and function in generally healthy, young adult black women who are vitamin D deficient or insufficient at baseline?
* Does 8 weeks of oral vitamin D3 supplementation (5,000 IU per day) improve various measures of laboratory blood pressure regulation and autonomic function?

All participants will undergo baseline testing, which includes 2 continuous weeks of objective sleep monitoring using a sleep watch, one 24-hour period of ambulatory blood pressure monitoring, and one blood vessel function testing visit. Following baseline testing, vitamin D insufficient and deficient participants will be prescribed take 5,000 IU of vitamin D3 daily for 8 continuous weeks. Participants will undergo 2-weeks of sleep monitoring again during weeks 3-4 of the supplementation period and during weeks 7-8 of the supplementation period. Additionally, 24-hour blood pressure monitoring will be performed during week 4 and week 8, and blood vessel function testing will take place at the end of week 4 and again at the end of week 8.

Researchers will assess the effect of the vitamin D3 supplementation intervention by comparing all values between baseline, week 4, and week 8 to see if there is any effect of vitamin D3 supplementation on 24-hour blood pressure, sleep duration and regularity, and blood vessel structure and function following 4 and 8 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Self-identified race is Black
* 18-30 years old
* Serum 25-hydroxyvitamin D concentration between 8-29.9 ng/ml determined at screening visit

Exclusion Criteria:

* Unwilling or unable to give consent
* Unwilling or unable to undergo a venous blood draw
* Diagnosed with any chronic diseases or conditions including cardiometabolic diseases, cardiorespiratory diseases, chronic mental or psychological illness, musculoskeletal diseases/conditions, autoimmune diseases, cancer, gastrointestinal/malabsorption disorders, hyper-/hypocalcemia, hyper-/hypoparathyroidism, hyper-/hypothyroidism, kidney disease, or a history of kidney stones
* Taking medication that may influence blood pressure or blood vessel function
* Diagnosed with a sleep disorder (e.g., insomnia, restless leg syndrome, sleep apnea), or are at high risk for a sleep disorder according to the ISI (score >14) or STOP-bang (score ≥3) questionnaires
* Currently taking medications or supplements that affect sleep (e.g., Ambien, sedatives, melatonin, etc.)
* Currently working night-shift work
* Resting blood pressure >130 or >80 mmHg
* BMI >30 kg/m2
* Currently pregnant, breast feeding, peri-menopausal, or post-menopausal
* Currently use tobacco (≥1 cigarette in the last month)
* Had COVID-19 in the past 60 days
* Received the COVID-19 vaccine or booster within in the past 14 days

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women assigned female at birth who currently identify as female
Enrollment: 22 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory systolic and diastolic blood pressure (mmHg) using an at-home ambulatory blood pressure monitor. | Change from baseline blood pressure values at 4 weeks and 8 weeks.
  Participants will undergo a 24-hour period of ambulatory systolic and diastolic blood pressure (mmHg) recording to evaluate diurnal systolic and diastolic blood pressure and nocturnal systolic and diastolic blood pressure.
Change in objectively estimated sleep duration and sleep efficiency using a Philips Actiwatch Spectrum Plus accelerometer wrist watch | Change from baseline sleep duration and sleep efficiency at 4 weeks and 8 weeks.
  Participants will undergo a two-week period of objectively estimated sleep recording using the Actiwatch. Sleep duration will be calculated as the average time spent asleep each night (hours) and sleep efficiency will be calculated as (total time asleep/total time in bed)*100%. Changes from baseline will be compared at week 4 and week 8.
Change in serum 25(OH)D concentration | Change from baseline 25(OH)D at 4 weeks and 8 weeks.
  Serum 25-hydroxyvitamin D concentration will be clinically assessed via Labcorp testing services.

SECONDARY OUTCOMES:
Change in brachial artery pulse wave analysis using the Sphygmocor XCEL system | Change in pulse wave analysis measures from baseline, week 4, and week 8
  Brachial systolic and diastolic blood pressure (BP) will be measured using the Sphygmocor XCEL system and central BP, augmentation index, and arterial wave reflections will be estimated via partial cuff inflation. Changes from baseline will be compared at week 4 and week 8.
Change in carotid-femoral pulse wave velocity using the Sphygmocor XCEL system (m/s) | Change in pulse wave velocity from baseline, week 4, and week 8
  Carotid to femoral pulse wave velocity (m/s) will be calculated using the Sphygmocor XCEL system. Changes from baseline will be compared at week 4 and week 8.
Change in ultrasound-assessed common carotid pulsatility index | Change in carotid pulsatility index from baseline, week 4, and week 8
  An duplex PW-mode image of the common carotid artery will be recorded for 20 heart cycles using ultrasonography. Blood velocity will be evaluated directly on the ultrasound and pulsatility index will be calculated for each cardiac waveform as peak systolic velocity - end diastolic velocity / mean velocity and averaged over 20 cardiac cycles. Changes from baseline will be compared at week 4 and week 8.
Change in ultrasound-assessed femoral artery blood flow response passive leg movement (PLM) (ml/min) | Change in femoral blood flow response to PLM from baseline, week 4, and week 8
  Femoral artery blood velocity and diameter will be continuously recorded using Doppler ultrasound for 1 minute at rest and during 1 minute of passive movement of the lower leg at the knee joint at a frequency of 1 hertz. Femoral artery blood flow will be calculated at baseline and during movement. The change in femoral artery blood flow will be calculated as peak blood flow during movement minus baseline blood flow. The change in femoral blood flow from baseline to peak is our assessment of femoral artery blood flow response to passive leg movement for which changes from baseline will be compared at week 4 and week 8.
Change in brachial artery flow-mediated dilation and reactive hyperemia | Change in FMD responses from baseline, week 4, and week 8
  Brachial artery reactivity will be assessed via the flow-mediated dilation technique and percent dilation of the brachial artery in response to 5 minutes of forearm arterial occlusion will be assessed offline via Medical Imaging Applications Brachial Analyzer software. Brachial artery blood velocity will be measured on the ultrasound as mean velocity throughout the test and blood flow will be calculated using arterial diameter. Brachial artery blood flow area under the curve and peak brachial artery blood flow following cuff release will be assessed at baseline, week 4, and week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Michele N D'Agata, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT05656742/ICF_001.pdf